CLINICAL TRIAL: NCT00728104
Title: Co-Enzyme Q10, L-Carnitine and Amitriptyline Usage in Cyclic Vomiting Syndrome (CVS): A Research Study
Brief Title: The Use of L-Carnitine And CoQ10 Supplements In the Treatment of Cyclic Vomiting Syndrome (CVS)
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, B Li, Professor of Pediatrics, MD, Medical College of Wisconsin
Other Study IDs: 090
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Cyclic Vomiting Syndrome
Keywords: Learn; L-Carnitine; Co-enzyme Q10; Effective; These supplements; Compared; Standard
MeSH Terms: conditions — Familial cyclic vomiting syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: The General Questionnaire: help to understand which characteristics of CVS patients are associated with both beneficial and harmful effects of these treatments
- 2: The Co-Enzyme Q10 Questionnaire: to be completed by individuals who ever taken co-enzyme Q10
- 3: The L-Carnitine Questionnaire: to be completed by individuals who have ever taken L-carnitine
- 4: The Amitriptyline Questionnaire: to be completed by individuals who have ever taken amitriptyline

SUMMARY:
This is a study with the principle goal being to learn about the use of L-Carnitine and CoQ10, two vitamin supplements that are currently being used to treat Cyclic Vomiting Syndrome, largely initiated by parents. We want to learn how effective these supplements are compared to standard treatment, at what dose, and what onset of action in order to initiate future prospective study on these supplements.

ELIGIBILITY:
Inclusion Criteria:

* 3 discrete episodes of vomiting
* normal health between episodes
* stereotypical clinical pattern
* no abnormal test results to account for vomiting (see exclusion criteria)

Exclusion Criteria:

* abnormal UGI with small bowel follow-through revealing an anatomic anomaly, inflammatory or obstructive
* Significantly abnormal endoscopic biopsies (moderate to severe esophagitis, H. pylori)
* Abnormal abdominal ultrasound revealing hydronephrosis, cholelithiasis, pancreatitis
* Positive screening for endocrine disorder (diabetic ketoacidosis, Addison's)
* Positive screening for inborn errors of metabolism (hypoglycemia, lactic acidosis, hyperammonemia, organic acidemia, amino aciduria, elevated beta-ALA, porphobilinogen)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cyclic Vomiting Syndrome (CVS) is a condition where children and adults have repeated attacks of severe vomiting, nausea, abdominal pain, headaches, and tiredness. These episodes can last from several hours to several days.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
How two vitamin supplements are being used to treat cyclic vomiting syndrome | Two years

SECONDARY OUTCOMES:
How effective these supplements appear to be compared to standard treatment | Two years

CONTACTS AND LOCATIONS:
Overall Officials: B Li, MD, Principal Investigator — Medical College of Wiconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- See also: Cyclic Vomiting Syndrome Association — http://www.cvsaonline.org